CLINICAL TRIAL: NCT02281461
Title: A Feasibility Study of PrePex Device for Infants and for Children, When Performed on Early Infants and Children Male Population by Physicians
Brief Title: Feasibility Study of PrePex Device When Performed on Early Infants & Children Male Population by Physicians
Acronym: RMC-06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Rwanda (Other Government)
Responsible Party: Principal Investigator, Vincent Mutabazi, Director of the Research Grants Unit, Ministry of Health, Rwanda
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RMC-06
Record Dates: First submitted 2014-10-05; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Medical Device Complication
Keywords: PrePex; Infants; Early infants; Children; Circumcision; HIV; AIDS; Non surgical
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early ifants (Experimental): Intervention Male circumcision using a non-surgical device
  Interventions: Device: Male circumcision using a non-surgical device
- Cildren (Experimental): Intervention Male circumcision using a non-surgical device
  Interventions: Device: Male circumcision using a non-surgical device

INTERVENTIONS:
Device: Male circumcision using a non-surgical device — Male Circumcision

SUMMARY:
The PrePex is a WHO prequalified medical device for adult male circumcision for HIV prevention. The Government of Rwanda was the first country to implement the PrePex and acts as the leading Center of Excellence providing training and formal guidelines.

In support of efforts to scale up male circumcision, readily available data have been applied to estimate the potential cost and impact of scaling up medical MC services in Rwanda to reach 80 percent of adult, children and newborn males by 2015. Infant and children male circumcision ensures that the wound will be healed before sexual activity begins, and thus reduces the risk of HIV transmission during healing period.

DETAILED DESCRIPTION:
The American Academy of Pediatrics (AAP) published in August 2012 a technical report and a policy statement, "Evaluation of current evidence indicates that the health benefits of new-born male circumcision outweigh the risks; furthermore, the benefits of newborn male circumcision justify access to this procedure for families who choose it. Specific benefits from male circumcision were identified for the prevention of urinary tract infections, acquisition of HIV, transmission of some sexually transmitted infections, and penile cancer. Male circumcision does not appear to adversely affect penile sexual function/sensitivity or sexual satisfaction. It is imperative that those providing circumcision are adequately trained and that both sterile techniques and effective pain management are used. Significant acute complications are rare."

The primary objective of the study was to assess the safety and efficacy of the PrePex device among healthy early infant and children males scheduled for voluntary circumcision. The study consisted of 2 phases:

Phase I included infants age 5-33 days Phase II included children age 4-10 years.

The study examined the feasibility of performing PrePex circumcision on early infants and children male population.

ELIGIBILITY:
Inclusion Criteria:

* Early infants and children males in ages - 5 to 33 days or 4-10 years
* Weighs more than 2500gr (for early infants)
* The infant or child should be healthy and in full-term
* Parent/legal guardian consent to the circumcision procedure
* Uncircumcised
* Parent/legal guardian able to understand the study procedures and requirements
* Parent/legal guardian agree to keep the infant for 48 hours or child for 24 hours hospitalization
* Parent/legal guardian agree to return to the health care facility for follow-up visits (or as instructed) after his circumcision until complete healing is achieved
* Parent/legal guardian able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have a good compliance for the study
* Parent/legal guardian agrees to anonymous video and photographs of the procedure and follow up visits.

Exclusion Criteria:

* Parent/legal guardian withhold consent
* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the participant from undergoing a circumcision
* Participant with the following diseases/conditions: Bilateral hydroceles, Curvature with penile torsion, Absence of ventral foreskin, Concealed penis (trapping urine beneath the foreskin), Megalourethra with deficiency of corpus spongiosum, Penoscrotal webbing, Epispadias, dorsal curvature, Hypospadias, Phimosis, paraphimosis, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias, epispadias, known haematological disorders and jaundice, yellow sclera or purpuric skin lesions, congenital abnormality
* Known bleeding / coagulation abnormality, uncontrolled diabetes
* Participant that to the opinion of the investigator is not a good candidate
* Parent/legal guardian does not agree to anonymous video and photographs of the procedure and follow up visits.

Ages: 5 Days to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of the PrePex device among early infants and children male population when performed by experienced surgeons | 2 weeks
  Safety by means of the following parameters: Moderate and Major Clinical adverse events and device-related incidents.

SECONDARY OUTCOMES:
Effectiveness of the PrePex device on early infants and children | 2 weeks
  Glans fully exposed (full circumcision)
Effectiveness of the PrePex device on early infants and children | 2 weeks
  Rate of foreskin dilations and adhesion separations
Effectiveness of the PrePex device on early infants and children | 2 weeks
  Time to device detachment
Effectiveness of the PrePex device on early infants and children | 2 weeks
  Time to complete healing
Effectiveness of the PrePex device on early infants and children | 2 weeks
  Rate of expected side effects
Effectiveness of the PrePex device on early infants and children | 2 weeks
  Rate of pain / discomfort
Effectiveness of the PrePex device on early infants and children | 2 weeks
  Rate of voiding

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul Bitega, M.D., Principal Investigator — Military Insurance, Medical Head of Clinical Affairs
Locations (1):
- Rwanda Military Hospital, Kigali, Kigali, Rwanda

REFERENCES:
- See also: Biomedical Center — http://www.rbc.gov.rw/